CLINICAL TRIAL: NCT05324540
Title: A First in Human Evaluation of a Novel Approach to Painless Cardioversion (NAPC) in Patients With Atrial Fibrillation
Acronym: NAPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MediCool Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FIH-001
Record Dates: First submitted 2022-03-18; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cool therapy (Experimental): A chilled instrument that has been chilled to a proscribed temperature will be applied to the oblique sinus. The instrument may be applied for up to 3 minutes per application and up to 3 times per patient.
  Interventions: Other: Cool therapy

INTERVENTIONS:
Other: Cool therapy — Application of cool therapy. A chilled (between 5C and 10C) instrument will be applied to the oblique sinus while the patient is in atrial fibrillation.

SUMMARY:
An assessment of the use of cold therapy to terminate atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years or older
* Male of female
* Subject has documented paroxysmal, or persistent atrial fibrillation (AF) with a history of less than one-year duration
* Must be in AF at time of surgery, or inducible using manual or electrical stimulation
* Subject is willing and able to provide written informed consent
* Subject has a life expectancy of at least 1 yearExclusion Criteria:

Exclusion Criteria: • Long-standing AF (duration > 1 year)

* Prior AF ablation
* Left main coronary artery occlusion > 70%
* Critical aortic stenosis (gradient > 50mm HG)
* Inability to induce patient into AF without drugs at time of surgery
* Female subjects who are pregnant at time of surgery
* Subjects with a medical condition or comorbidity that could adversely impact study participation, safety or conduct of the study
* Permanent pacemaker or implantable cardioverter defibrillator
* Current cancer treatment that includes radiation of the heart
* Inability to give informed consent
* Significant intra-cardiac thrombus
* Subjects not eligible for or considered high risk for anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Termination of atrial fibrillation | Termination will be measured within 3 minutes of application of cool therapy. No longer term data will be collected.
  Number of successful terminations of atrial fibrillation to normal sinus rhythm upon application of cool therapy will be measured and assessed.

SECONDARY OUTCOMES:
Time to termination | Time to termination will be assessed only during each application. No longer term data will be collected.
  The time it takes (in minutes and seconds) to terminate atrial fibrillation to normal sinus rhythm will be measured following application of cool therapy.

IPD SHARING:
Plan to Share IPD: No